CLINICAL TRIAL: NCT02260401
Title: Long Term Outcomes of Lumbar Epidural Steroid Injections for Spinal Stenosis
Acronym: LESSER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Janna Friedly, Assistant Professor, Rehabilitation Medicine, University of Washington
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 39023
Record Dates: First submitted 2014-10-05; First posted 2014-10-09 (Estimated); Results first posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-03

CONDITIONS: Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Individualized report (Experimental): Each patient in this group will receive an individualized report with their own outcome data (pain and function) during the first year of the LESS trial. They will receive these reports at 18 months.
  Interventions: Other: Individualized report
- Individualized Reports after 24 months (No Intervention): Patients in this group will receive the individualized report, but will not receive it until after the conclusion of the study at 24 months. They will serve as the control group.

INTERVENTIONS:
Other: Individualized report — Each patient will receive an individualized report that contains their own outcome data for the first years of the LESS trial (including pain and function following treatment with epidural injections)
  Arms: Individualized report

SUMMARY:
Spinal stenosis is one of the most common causes of low back pain among older adults and can result in significant disability. Despite this, it still isn't known which treatments are most effective or what outcomes are most important to these older adults. Through a Patient Centered Outcomes Research Institute (PCORI) contract, the investigators are building on the existing infrastructure of an AHRQ-funded (ARRA CHOICE award) comparative effectiveness research (CER) trial of epidural steroid injections (ESI) for spinal stenosis (the LESS trial) to address several critical research questions. The proposed study will answer the following key questions. Do decision aids tailored to older adults with spinal stenosis change patient decision-making regarding subsequent treatments? Do patients respond differently at subsequent outcome assessments time-points after receiving tailored decision aids that contain their own individual outcome data from prior treatments? The investigators hypothesize that providing these individualized reports will allow patients to make more informed choices regarding subsequent treatments, leading to reduced use of ineffective treatments and improved outcomes overall.

DETAILED DESCRIPTION:
LESS trial participants will be randomized to receive the individualized outcome report before the 18-month interview or after the 24-month follow up. Both groups will be asked to rank outcome domains of most importance to them, to answer questions regarding their beliefs about receiving future treatments for spinal stenosis and to complete the standard self-reported outcomes questionnaire. In addition, we will ask the study participants whether the information presented in the individualized report was helpful in deciding their future epidural injection treatments as well as if the content of the reports was easy to understand. At 24 months, we will repeat the interview and the outcomes assessment. We will again compare the groups in terms of their responses to determine if there are lasting differences in how patients who received the individualized reports make decisions regarding future treatments and respond to the self-reported outcomes questions. In addition, we will compare healthcare utilization between the two groups from 18 months to 24 months to determine if providing the individualized outcomes reports changed treatment utilization (i.e., do people who receive the report undergo fewer subsequent injections or other treatments for pain?). We hypothesize that providing these individualized reports will allow patients to make more informed choices regarding subsequent treatments, leading to reduced use of ineffective treatments and improved outcomes overall.

ELIGIBILITY:
Inclusion Criteria:

Patients already enrolled in the LESS trial will be eligible for participation in the LESSER trial

Exclusion Criteria:

none

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2013-10; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Individualized Report | Individualized Reports After 24 Months
Started | 80 | 85
Completed | 75 | 73
Not Completed | 5 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Individualized Report | Individualized Reports After 24 Months | Total
Number analyzed (Participants) | 80 | 85 | 165
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (10) | 69.1 (9.4) | 67.8 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 43 | 79
  Male | 44 | 42 | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 75 | 81 | 156
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Utilization of ESI
Description: We will measure whether or not providing these individualized reports to patients impacts patients decision-making regarding use of epidural steroid injections between 18 and 24 months
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: number of ESI between 18-24 months
Arm/Group | Individualized Report | Individualized Reports After 24 Months
Number analyzed (Participants) | 80 | 85
number of ESI between 18-24 months | 3.6 (2.0) | 3.3 (2.0)

2. Secondary Outcome: Healthcare Utilization
Description: We will determine if providing individualized reports to the LESS trial participants at 198 months impacts healthcare utilization for spinal stenosis between 18 and 24 months (including doctors visits, physical therapy, surgery, opioid use)
Time Frame: 24 months
Reporting Status: Not Posted, anticipated posting 2017-04

ADVERSE EVENTS:
Arm/Group | Individualized Report | Individualized Reports After 24 Months
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/85
Other Adverse Events (participants affected / at risk) | 0/80 | 0/85

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No